CLINICAL TRIAL: NCT03163459
Title: Short-duration Selective Brain Cooling for Ischemic Stroke Patients Undergoing Mechanical Thrombectomy: a Randomized Controlled Trial
Brief Title: Short-duration Selective Brain Cooling for Patients Undergoing Mechanical Thrombectomy
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Interim analysis
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Vice President, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ET-EH
Record Dates: First submitted 2017-05-06; First posted 2017-05-23 (Actual); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Hypothermia; Stroke, Acute
Keywords: mechanical thrombectomy; selective brain cooling
MeSH Terms: conditions — Hypothermia; Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mechanical thrombectomy group (Active Comparator): Conventional mechanical thrombectomy
  Interventions: Device: mechanical thrombectomy
- mechanical thrombectomy plus selective brain cooling group (Experimental): A microcatheter which was used to deploy the stent retriever was threaded into the femoral artery in the groin through a guiding catheter and up through the neck, until it reached beyond the clot causing the stroke under the assistance of micro-guide wire, 50 mL cold 0.9% saline (4°C) was infused into the ischemic territory at 10 mL/min through the microcatheter, thus allowing the cold solution to infuse into the ischemic territory prior to reperfusion. After that, mechanical thrombectomy with a stent retriever was performed to recanalize the occluded vessel as soon as possible. After the recanalization, cold 0.9% saline (4°C) was infused into the ischemic brain tissue through the guide catheter at 30 mL/min for 10 minutes.
  Interventions: Drug: selective brain cooling by cold saline perfusion; Device: mechanical thrombectomy

INTERVENTIONS:
Drug: selective brain cooling by cold saline perfusion — During the procedure, a microcatheter which was used to deploy the stent retriever was threaded into the femoral artery in the groin through a guiding catheter and up through the neck, until it reached beyond the clot causing the stroke under the assistance of micro-guide wire, 50 mL cold 0.9% saline (4°C) was infused into the ischemic territory at 10 mL/min through the microcatheter, thus allowing the cold solution to infuse into the ischemic territory prior to reperfusion. After that, mechanical thrombectomy with a stent retriever was performed to recanalize the occluded vessel as soon as possible. After the recanalization, cold 0.9% saline (4°C) was infused into the ischemic brain tissue through the guide catheter at 30 mL/min for 10 minutes.
  Arms: mechanical thrombectomy plus selective brain cooling group
Device: mechanical thrombectomy — conventional mechanical thrombectomy using Solitaire

SUMMARY:
To determine the efficacy and safety of short-duration intra-artery selective brain cooling in addition to mechanical thrombectomy in patients with acute ischemic stroke.

DETAILED DESCRIPTION:
Acute ischemic stroke remains one of the leading causes of disability and death in both developed and developing countries. Using intravenous thrombolysis combined with intra-arterial therapy to recanalize occluded vessels in eligible patients is recommended by current guidelines. Five randomized clinical trials showed that modified thrombolysis in cerebral ischemia (mTICI) 2b/3 recanalization can be achieved in 59-88% of acute ischemic stroke patients with anterior circulation large artery occlusion，but only an average of 46% of patients have a favorable outcome (modified Rankin Scale score [mRS] 0-2). Therefore, new therapeutic strategies in addition to thrombectomy for acute ischemic stroke are urgently needed.

As early as 1987, Busto et al. found that lowering of the brain temperature by only a few degrees during ischemia confers a marked neuroprotective effect. Therapeutic hypothermia has been suggested to be the most potent neuroprotective strategy in recent years5，and a number of clinical studies in patients with acute cerebral infarction also showed that mild hypothermia (33-35 ℃) can increase tolerance to ischemic insults and play a significant neuroprotective role after reperfusion. However, adverse events such as pneumonia, affecting up to 35% of treated patients occurs with hypothermia. Since selective brain cooling does not require a reduction in core body temperature, it is theoretically possible to avoid many serious adverse effects caused by whole body hypothermia.

The investigators have previous shown that short-duration selective brain cooling by the intra-arterial infusion of cold saline combined with mechanical thrombectomy in acute ischemic stroke is feasible and safe. The efficacy of selective brain cooling in patients undergoing mechanical thrombectomy, however, is not established. The investigators therefore conducted this RCT study to explore the efficacy of short-duration selective brain cooling in patients with acute ischemic stroke who underwent mechanical thrombectomy.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke within 6 hours from symptom onset/last seen well.
* Occlusion (TIMI 0-1) of the basilar artery or distal intracranial carotid artery or middle (M1/M2) or anterior (A1/A2) cerebral artery as evidenced by CTA/MRA/DSA.
* Age ≥18 and ≤80
* No significant pre-stroke functional disability (mRS ≤ 1)
* The possibility to start treatment within 6 hours from onset.
* Informed consent given

Exclusion Criteria:

* Known hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with INR > 3.0
* Baseline platelet count < 50.000/µL
* Baseline blood glucose of < 50mg/dL or >400mg/dl
* Severe, sustained hypertension (SBP > 220 mm Hg or DBP > 110 mm Hg) NOTE: If the blood pressure can be successfully reduced and maintained below these levels using commonly used medications in China for these purposes (including iv antihypertensive drips), the patient can be enrolled.
* Serious, advanced, or terminal illness with anticipated life expectancy of less than one year.
* History of life threatening allergy (more than rash) to contrast medium
* Subjects who has received iv t-PA treatment beyond 4.5 hours from the beginning of the symptoms.
* Patients with acute stroke within the first 48 hours after percutaneous cardiac, cerebrovascular interventions and major surgery
* Renal insufficiency with creatinine ≥ 3 mg/dl
* Woman of childbearing potential who is known to be pregnant or lactating or who has a positive pregnancy test on admission.
* Subject participating in a study involving an investigational drug or device that would impact this study.
* Cerebral vasculitis
* Patients with a pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations, mRS score at baseline must be ≤ 1, which includes patients who are severely demented, require constant assistance in a nursing home type setting or who live at home but are not fully independent in activities of daily living (toileting, dressing, eating, cooking and preparing meals, etc.)
* Unlikely to be available for 90 days follow-up (e.g. no fixed home address, visitor from overseas).
* CT or MR evidence of hemorrhage (the presence of microbleeds on MRI is allowed).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-02-06 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-12-16 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieving favorable outcomes defined as mRS 0-2 at 90 days as evaluated by independent central assessors who are blinded to treatment | 90 days
  mRS 0-2

SECONDARY OUTCOMES:
Dramatic early favorable response | 24 hours
  an NIHSS of 0-2 or NIHSS improvement ≥ 8 points at 24 (-2/+12 hours) hours from randomization or before discharge if patient is discharged prior to the above time limit
Final infarct volume evaluated on CT/MR at 24 hours (-2/+12 hours) | 24 hours
  Final infarct volume evaluated on CT/MR at 24 hours (-2/+12 hours)
The change of infarct volume compared with baseline. | 24 hours
  The change of infarct volume compared with baseline.
Vessel recanalization | 24 hours
  Vessel recanalization evaluated by angiography (one of CT angiography , MR Angiography and conventional angiography) at 24 hours (-2/+12 hours) in both treatment groups
Barthel Index at 90 days | 90 days
  Barthel Index at 90 days
NIHSS at 90 days | 90 days
  NIHSS at 90 days
Proportion of patients achieving excellent favorable outcomes defined as mRS 0-1 at 90 days | 90 days
  mRS 0-1 at 90 days
mRS shift analysis at 90 days | 90 days
  mRS shift analysis

OTHER OUTCOMES:
Mortality at 90 days | 90 days
  Mortality
Clinically significant ICH rates at 24 (-2/+12) hours. | 24 hours
  All intracerebral hemorrhages will be classified by a central core-lab using the Heidelberg criteria. Symptomatic ICH will be defined as per the SITS-MOST definition: deterioration in NIHSS score of ≥4 points within 24 hours from treatment and evidence of intraparenchymal hemorrhage type 2 in the 22 to 36 hours follow-up imaging scans. The incidence of any asymptomatic hemorrhage measured at 24 (-2/+12) hours will also be compared
Procedural related complications | From the operation to 24 hours after the operation
  arterial perforation, arterial dissection, and embolization in a previously uninvolved vascular territory
Rectal temperature | From 1 hour before operation to 1 hours after operation
  Rectal temperature
Hematocrit | From 3 hour before operation to 3 hours after operation
  Hematocrit
blood biochemistry | From 3 hour before operation to 3 hours after operation
  Routine blood test and blood biochemistry
Vital signs | From 1 hour before operation to 24 hours after operation
  Vital signs

CONTACTS AND LOCATIONS:
Locations (1):
- Xuan Wu Hospital，Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen J, Liu L, Zhang H, Geng X, Jiao L, Li G, Coutinho JM, Ding Y, Liebeskind DS, Ji X. Endovascular Hypothermia in Acute Ischemic Stroke: Pilot Study of Selective Intra-Arterial Cold Saline Infusion. Stroke. 2016 Jul;47(7):1933-5. doi: 10.1161/STROKEAHA.116.012727. Epub 2016 May 19. PMID 27197848